CLINICAL TRIAL: NCT01100437
Title: A Single-Center, Randomized, Double-Blind, Two-Way Crossover Study to Evaluate Whether a Single-Dose Administration of Crushed and Whole EMBEDA Induces Clinical Opiate Withdrawal Signs and Symptoms in Opioid-Dependent Patients With Chronic, Non-Cancer Pain Who Are Stabilized on EMBEDA¿
Brief Title: Safety Study to Assess Opiate Withdrawal Signs and Symptoms in Opioid Dependent Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: ALO-01-09-111; B4541002
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Results first posted 2012-03-28 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Pain
Keywords: opioid; morphine; naltrexone; withdrawal signs; withdrawal symptoms
MeSH Terms: conditions — Chronic Pain; Substance Withdrawal Syndrome | interventions — morphine, naltrexone combination; Morphine; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMBEDA™ (morphine sulfate/naltrexone hydrochloride) crush (Experimental): EMBEDA (morphine sulfate plus naltrexone hydrochloride ER) capsules crushed and mixed in solution and administered orally at each patient's stable dose, given either once daily or twice daily.
  Interventions: Drug: EMBEDA™ (morphine sulfate/naltrexone hydrochloride) crush
- EMBEDA™ (morphine sulfate/naltrexone hydrochloride) whole (Experimental): EMBEDA (morphine sulfate plus naltrexone hydrochloride ER) capsules, administered orally and intact at each patient's stable dose, given either once daily or twice daily
  Interventions: Drug: EMBEDA™ (morphine sulfate/naltrexone hydrochloride) whole

INTERVENTIONS:
Drug: EMBEDA™ (morphine sulfate/naltrexone hydrochloride) crush — Placebo capsules plus EMBEDA capsules crushed and mixed in solution administered orally at each patient's stable dose, given either once daily or twice daily
  Arms: EMBEDA™ (morphine sulfate/naltrexone hydrochloride) crush
Drug: EMBEDA™ (morphine sulfate/naltrexone hydrochloride) whole — EMBEDA capsules, administered orally and intact at each patient's stable dose, given either once daily or twice daily with 150mL placebo solution
  Arms: EMBEDA™ (morphine sulfate/naltrexone hydrochloride) whole

SUMMARY:
This study will evaluate whether crushed EMBEDA capsules induce clinical opiate withdrawal signs and symptoms in opioid-dependent patients with chronic non-cancer pain who are stabilized on EMBEDA.

DETAILED DESCRIPTION:
The decision to terminate the trial was due to a lack of study drug supply. Decision was not based on any safety concerns. The date of the notification of termination letter was March 11, 2011.

ELIGIBILITY:
Inclusion Criteria:

* Chronic moderate to severe non-cancer pain that has been treated with opioid analgesics for at least three months (with stabilized pain control and stabilized dose for 28 days prior to enrollment).
* Receiving an opioid dose equivalent to 20 mg - 120 mg morphine once or twice daily.
* Patient displays signs and symptoms of withdrawal (i.e., COWS score ≥5) following naloxone administration during the Naloxone Challenge.

If female and able to become pregnant, must use an approved method of birth control.

* Excluding the chronic moderate to severe non-cancer pain, the patient is judged by the Investigator to be in generally good health at screening based upon the results of a medical history, physical examination, laboratory profile, and 12 lead electrocardiogram (ECG).

Exclusion Criteria:

* Female who is pregnant or breastfeeding.
* Patient has a known allergy or history of significant adverse reaction to morphine, other opioids, naltrexone, acetaminophen, or related compounds.
* Patient is receiving systemic chemotherapy, has an active malignancy of any type, or has been diagnosed with cancer within the 5 years prior to screening (excluding squamous or basal cell carcinoma of the skin).
* History of, or ongoing, alcohol or drug abuse.
* Patient has made a donation of blood or has had a significant blood loss within 30 days prior to screening.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Setnik B, Roland CL, Goli V, Sommerville K, Webster L. A clinical trial to determine if corelease of morphine and naltrexone from crushed extended-release capsules induces withdrawal in opioid-dependent patients: a descriptive analysis of six patients. J Opioid Manag. 2013 Mar-Apr;9(2):139-50. doi: 10.5055/jom.2013.0155. PMID 23709323
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=ALO-01-09-111&StudyName=Safety%20Study%20to%20Assess%20Opiate%20Withdrawal%20Signs%20and%20Symptoms%20in%20Opioid%20Dependent%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- EMBEDA Capsule Then EMBEDA Solution: EMBEDA (morphine sulfate plus naltrexone hydrochloride) Extended Release (ER) capsule(s) were administered orally once or twice a day (20 milligrams [mg] to 120 mg). During the open label titration and stabilization phase EMBEDA was administered and titrated to a dose that adequately managed the participants pain up to 35 days. In the open label Maintenance Phase the participant was administered the established stable dose for a minimum of 7 days up to 28 days. The participant was then randomized to one of two double-blind treatment sequences for the Treatment Phase. During the Treatment Phase the participant was administered whole EMBEDA capsules orally at participant's stable dose along with a matched placebo solution in the first intervention period. In the second intervention period the participant received crushed EMBEDA capsules that were mixed in solution and administered orally at participant's stable dose along with matched placebo capsules.
- EMBEDA Solution Then EMBEDA Capsule: EMBEDA (morphine sulfate plus naltrexone hydrochloride) ER capsule(s) were administered orally once or twice a day (20 mg to 120 mg). During the open label titration and stabilization phase EMBEDA was administered and titrated to a dose that adequately managed the participants pain up to 35 days. In the open label Maintenance Phase the participants were administered the established stable dose for a minimum of 7 days up to 28 days. The participant was then randomized to one of two double-blind treatment sequences for the Treatment Phase. During the Treatment Phase the participant was administered crushed EMBEDA capsules orally at participants stable dose mixed in solution along with matched placebo capsules in the first intervention period. In the second intervention period the participant received whole EMBEDA capsules administered orally at participant's stable dose along with matched placebo solution.
- EMBEDA Capsule: EMBEDA (morphine sulfate plus naltrexone hydrochloride) ER capsule(s) were administered orally once or twice a day (20 mg to 120 mg). During the titration and stabilization phase EMBEDA was administrated and titrated to a dose that adequately managed the participants pain for up to 35 days. In the Maintenance Phase the participant's were administered the established stable dose for a minimum of 7 days up to 28 days. Participants were not randomized to treatment phase.
Period: Screening
Arm/Group | EMBEDA Capsule Then EMBEDA Solution | EMBEDA Solution Then EMBEDA Capsule | EMBEDA Capsule
Started | 4 | 2 | 8
Completed | 4 | 2 | 8
Not Completed | 0 | 0 | 0
Period: Titration/Stabilization
Arm/Group | EMBEDA Capsule Then EMBEDA Solution | EMBEDA Solution Then EMBEDA Capsule | EMBEDA Capsule
Started | 4 | 2 | 8
Completed | 4 | 2 | 2
Not Completed | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Non-compliance | 0 | 0 | 1
Not completed — Sponsor canceled study | 0 | 0 | 1
Period: Maintenance
Arm/Group | EMBEDA Capsule Then EMBEDA Solution | EMBEDA Solution Then EMBEDA Capsule | EMBEDA Capsule
Started | 4 | 2 | 2
Completed | 4 | 2 | 0
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Sponsor termination of study | 0 | 0 | 1
Period: Treatment 1
Arm/Group | EMBEDA Capsule Then EMBEDA Solution | EMBEDA Solution Then EMBEDA Capsule | EMBEDA Capsule
Started | 4 | 2 | 0
Completed | 4 | 2 | 0
Not Completed | 0 | 0 | 0
Period: Washout (4 Days)
Arm/Group | EMBEDA Capsule Then EMBEDA Solution | EMBEDA Solution Then EMBEDA Capsule | EMBEDA Capsule
Started | 4 | 2 | 0
Completed | 4 | 2 | 0
Not Completed | 0 | 0 | 0
Period: Treatment 2
Arm/Group | EMBEDA Capsule Then EMBEDA Solution | EMBEDA Solution Then EMBEDA Capsule | EMBEDA Capsule
Started | 4 | 2 | 0
Completed | 4 | 2 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: EMBEDA (morphine sulfate plus naltrexone hydrochloride) ER capsule(s) were administered orally once or twice a day (20 mg to 120 mg). During the titration and stabilization phase EMBEDA was administered and titrated to a dose that adequately managed the participant's pain up to 35 days. The participants then started the Maintenance Phase and were administered the established stable dose of EMBEDA for a minimum of 7 days up to 28 days. Eligible participants were randomized into the 2 treatment groups.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 14
Age Continuous [Median (Full Range); unit: years] | 45.2 [32.6 to 67.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Opiate Withdrawal Scale (COWS) Score Greater Than or Equal to (≥) 13 in the Treatment Phase
Description: COWS is an 11 section clinical assessment of withdrawal symptoms, each section is rated from 0 (no symptom) to 4 or 5 (most severe symptom). Total score is classified into a 4 point rating scale (mild 5-12, moderate 13-24, moderately severe 25-36 and severe more than 36 points).
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24 hours (hr) post-dose and unscheduled assessment (UA)
Population: Intent-to-treat population (ITT): all randomized participants who received at least one dose of double-blind treatment in the Treatment Phase and had at least one post-dose pharmacodynamic assessment completed in the Treatment Phase.
Measure: Number; unit: participants
Groups:
- EMBEDA Whole Capsules: EMBEDA whole capsules, administered orally at participant's stable dose (20 mg to 120 mg), given once or twice daily along with matched placebo solution in any treatment period.
- EMBEDA Crushed in Solution: EMBEDA capsules crushed mixed in solution and administered orally at participant's stable dose (20 mg to 120 mg), given once or twice daily with matched placebo whole capsules in any treatment period.
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 6 | 6
participants | 1 | 3

2. Secondary Outcome: Average Numeric Pain Rating Scale (NPRS) in Titration/Stabilization and Maintenance Phases
Description: Average pain scores in the previous 24 hours using an 11 point NPRS ranging from no pain (0) to worst pain (10).
Time Frame: Baseline up to Day 63
Population: ITT; N=number of participants with evaluable data; n=number of participants evaluated at the specific time point
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EMBEDA Capsules: EMBEDA whole capsules, administered orally at participant's stable dose (20 mg to 120 mg), given once or twice daily along with matched placebo solution in any treatment period.
Arm/Group | EMBEDA Capsules
Number analyzed (Participants) | 6
units on a scale
  Titration/Stabilization-Baseline (n=6) | 5.5 (1.05)
  Titration/Stabilization-Visit 2b (n=6) | 5.2 (2.23)
  Titration/Stabilization-Visit 2c (n=2) | 5.5 (3.54)
  Titration/Stabilization-Visit 2d (n=1) | 3.0 (NA) — Not applicable (NA). One participant with analyzable data, no standard deviation calculated.
  Maintenance (n=6) | 4.2 (1.94)

3. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) During the Treatment Phase
Description: Average Tmax for Morphine, Naltrexone and 6-β-Naltrexol
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: Pharmacokinetic (PK) population: all randomized participants who received at least one dose of EMBEDA (whole or crushed) in the Treatment Phase and had at least one PK assessment completed in the Treatment Phase; n=number of participants with evaluable data for the specific category
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 6 | 6
hours (h)
  Morphine (n=6,6) | 5.67 (2.658) | 1.29 (0.813)
  Naltrexone (n=0,6) | NA (NA) — No participants with evaluable data | 1.46 (0.697)
  6-β-Naltrexol (n=4,6) | 6.13 (11.919) | 1.63 (0.787)

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) During the Treatment Phase
Description: Average Cmax for Morphine, Naltrexone and 6-β-Naltrexol
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: PK population; n=number of participants with evaluable data for specific category
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 6 | 6
nanogram per milliliter (ng/mL)
  Morphine (n=6,6) | 27.5 (14.14) | 70.4 (47.88)
  Naltrexone (n=0,6) | NA (NA) — No participants with evaluable data | 321.1 (225.05)
  6-β-Naltrexol (n=4,6) | 24.4 (15.40) | 3398.3 (1327.97)

5. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) During the Treatment Phase
Description: Average Cmin for Morphine, Naltrexone and 6-β-Naltrexol
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: PK population; n=number of participants with evaluable data for specific category
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 6 | 6
ng/mL
  Morphine (n=6,6) | 13.8 (6.89) | 11.2 (8.86)
  Naltrexone (n=0,6) | NA (NA) — No participants with evaluable data | 6.9 (1.17)
  6-β-Naltrexol (n=4,6) | 15.9 (9.29) | 42.7 (66.93)

6. Secondary Outcome: Apparent Oral Clearance (CL/F) During the Treatment Phase
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: PK population; N=number of participants with evaluable data; n=number of participants with evaluable data for the specific category
Measure: Mean (Standard Deviation); unit: liters/hour (L/h)
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 3 | 6
liters/hour (L/h)
  Morphine (n=2,6) | 37.6 (11.53) | 77.2 (25.36)
  Naltrexone (n=0,6) | NA (NA) — No participants with evaluable data | 75151.0 (51706.48)
  6-β-Naltrexol (n=3,6) | 45143.6 (14157.49) | 1758.0 (381.67)

7. Secondary Outcome: Volume of Distribution (Vd/F)During the Treatment Phase
Description: Average Vd/F for Morphine, Naltrexone and 6-β-Naltrexol
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: PK population; N=number of participants with evaluable data; n=number of participants with evaluable date for the specific category
Measure: Mean (Standard Deviation); unit: liter (L)
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 3 | 6
liter (L)
  Morphine (n=2,6) | 3173.1 (1724.61) | 1668.2 (830.08)
  Naltrexone (n=0,6) | NA (NA) — No participants with evaluable data. | 304171.8 (206998.86)
  6-β-Naltrexol (n=3,6) | 3447244.4 (1868128.43) | 26304.5 (10730.59)

8. Secondary Outcome: Plasma Decay Half-Life (t1/2) During the Treatment Phase
Description: Average plasma decay half-life of morphine, naltrexone and 6-β-Naltrexol. Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 3 | 6
h
  Morphine (n=2,6) | 56.2 (14.55) | 17.0 (10.99)
  Naltrexone (n=0,6) | NA (NA) — No participants with evaluable data | 3.0 (1.10)
  6-β-Naltrexol (n=3,6) | 50.9 (11.77) | 10.1 (2.43)

9. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUC0-τ) During the Treatment Phase
Description: Average AUC0-τ for Morphine, Naltrexone and 6-β-Naltrexol reported. τ=24 hours
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: PK population; n=number of participants with evaluable data for the specific category
Measure: Mean (Standard Deviation); unit: ng times h divided by mL (ng*h/mL)
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 6 | 6
ng times h divided by mL (ng*h/mL)
  Morphine (n=6,6) | 513.4 (310.87) | 542.6 (366.62)
  Naltrexone (n=0,6) | NA (NA) — No participants with evaluable data | 1314.7 (1119.25)
  6-β-Naltrexol (n=4,6) | 463.5 (290.94) | 28891.2 (14871.70)

10. Secondary Outcome: Area Under the Curve From Time Zero to the Time of Last Measurable Concentration (AUC0-last) During the Treatment Phase
Description: Average AUC0-last for Morphine, Naltrexone and 6-β-Naltrexol. Area under the plasma concentration time-curve from time zero to the last measured concentration.
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: PK population; n=number of participants with evaluable data for the specific category
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 6 | 6
ng*h/mL
  Morphine (n=6,6) | 513.4 (310.87) | 542.6 (366.62)
  Naltrexone (n=0,6) | NA (NA) — No participants with evaluable data | 1300.0 (1131.24)
  6-β-Naltrexol (n=4,6) | 450.3 (312.56) | 28891.2 (14871.69)

11. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] During the Treatment Phase
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). Average AUC 0-∞ for Morphine, Naltrexone and 6-β-Naltrexol reported.
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 3 | 6
ng*h/mL
  Morphine (n=2,6) | 2023.5 (1935.01) | 887.7 (583.83)
  Naltrexone (n=0,6) | NA (NA) — No participants with evaluable data | 1330.7 (1141.75)
  6-β-Naltrexol (n=3,6) | 1469.5 (955.52) | 35297.8 (18407.20)

12. Other Pre Specified Outcome: Time to First Occurrence of a COWS Score ≥ 13 for Each Treatment During the Treatment Phase
Description: Average time to first occurrence of a COWS score ≥ 13
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24 hr post-dose and UA
Population: ITT; Subset of participants with COWS >= 13
Measure: Mean (Standard Error); unit: h
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 1 | 3
h | 2.5 (NA) — One participant with analyzable data, no standard error calculated. | 0.7 (0.02)

13. Other Pre Specified Outcome: Morphine Plasma Concentration at First COWS ≥ 13 in the Treatment Phase
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: ITT; Subset of participants with COWS ≥ 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 1 | 3
ng/mL | 16.00 (NA) — One participant with analyzable data, no standard deviation calculated. | 86.30 (53.316)

14. Other Pre Specified Outcome: Naltrexone Plasma Concentration at First COWS ≥ 13 in the Treatment Phase
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: ITT; Subset of participants with COWS ≥ 13
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 1 | 3
picogram/milliliter (pg/mL) | NA (NA) — No participants with evaluable data. | 350.50 (195.869)

15. Other Pre Specified Outcome: 6-β-Naltrexone Plasma Concentration at First COWS ≥ 13 in Treatment Phase
Time Frame: Prior to dose, 0, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, and 24 hr post-dose
Population: ITT; Subset of all participants with COWS ≥ 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 1 | 3
pg/mL | NA (NA) — No participants with evaluable data | 3375.00 (827.315)

16. Other Pre Specified Outcome: Maximum Post-dose COWS in the Treatment Phase
Description: as for outcome 1
Time Frame: Between 0.5 and 24 hours post-dose
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EMBEDA Whole Capsules | EMBEDA Crushed in Solution
Number analyzed (Participants) | 6 | 6
units on a scale | 3.7 (4.63) | 10.7 (6.83)

ADVERSE EVENTS:
Time Frame: Study procedure related adverse events (AEs) were collected from the time of written Informed Consent and all other AEs from the time of the first dose of EMBEDA at Visit 2.
Description: The same event may appear as both an AE and a serious adverse events (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- EMBEDA Whole Capsule Treatment Period: EMBEDA whole capsules, administered orally at participant's stable dose (20 mg to 120 mg), given once or twice daily along with matched placebo solution in any treatment period.
- EMBEDA Crushed in Solution Treatment Period: EMBEDA capsules crushed mixed in solution and administered orally at participant's stable dose (20 mg to 120 mg), given once or twice daily along with matched placebo whole capsules in any treatment period .
- EMBEDA Capsule Titration/Stabilization Period: EMBEDA capsule(s) administered orally once or twice a day (20 mg go 120 mg) to adequately manage the participants pain.
- EMBEDA Capsules Maintenance Period: EMBEDA capsule(s) administered orally once or twice a day dose (20 mg go 120 mg) at the participants stable dose for 7 days minimum.
Arm/Group | EMBEDA Whole Capsule Treatment Period | EMBEDA Crushed in Solution Treatment Period | EMBEDA Capsule Titration/Stabilization Period | EMBEDA Capsules Maintenance Period
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 4/6 | 6/6 | 12/14 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EMBEDA Whole Capsule Treatment Period (N=6) | EMBEDA Crushed in Solution Treatment Period (N=6) | EMBEDA Capsule Titration/Stabilization Period (N=14) | EMBEDA Capsules Maintenance Period (N=8)
Headache (Nervous system disorders) | 3 | 3 | 0 | 0
Tremor (Nervous system disorders) | 1 | 4 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 6 | 6 | 0
Restlessness (Psychiatric disorders) | 1 | 3 | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Irritability (General disorders) | 1 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 1 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 2 | 3 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 2 | 1 | 0
Mydriasis (Eye disorders) | 0 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 5 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 2 | 0
Euphoric mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Sponsor terminated study early on 10-Mar-2011.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.